CLINICAL TRIAL: NCT04424888
Title: Evaluating Use of Continuous Glucose Monitors in a Short-term 2x2-Crossover Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pendulum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WB01-205
Record Dates: First submitted 2020-05-27; First posted 2020-06-11 (Actual); Results first posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Type 2; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- WB-011 (Experimental): 3 capsules administered twice daily with morning and evening meal for 2 weeks
  Interventions: Other: WB-011; Device: Continuous Glucose Monitor
- Placebo (Placebo Comparator): 3 capsules administered twice daily with morning and evening meal for 2 weeks
  Interventions: Other: Placebo; Device: Continuous Glucose Monitor

INTERVENTIONS:
Other: WB-011 — WB-011 medical food product.
  Arms: WB-011
Other: Placebo — Placebo Capsules identical to those containing WB-011.
  Arms: Placebo
Device: Continuous Glucose Monitor — Abbott Freestyle Libre(™) Glucose Sensors were used throughout the study.

SUMMARY:
This 5-week, double-blind, placebo-controlled, 2x2 crossover pilot study investigate the potential of collecting robust, real-time clinical study measures of glucose levels using Abbott Freestyle Libre Continuous Glucose Monitoring devices associated with a smartphone application

DETAILED DESCRIPTION:
The goal of this study is to characterize the performance of a Continuous Glucose Monitoring System in medical food studies. The Freestyle Libre Glucose Sensors will be used to follow subject's 8-day glucose trajectories over the course of a 5-week, double-blind, placebo-controlled, 2x2 crossover, medical-food experiment. The medical food has been designed to increase butyrate production and promote the health of the colonic mucin layer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years of age
* If female, must meet all the following criteria:
* Not pregnant or breastfeeding
* If of childbearing potential (including peri-menopausal women who have had a menstrual period within one year) must practice and be willing to continue to practice appropriate birth control (defined as a method which results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as double barrier methods [male condom with spermicide, with or without cervical cap or diaphragm], implants, injectable or oral contraceptives [must have been using for at least the last 3 months], some intrauterine contraceptive devices, tubal ligation, or in an established relationship with a vasectomized partner) during the entire duration of the study
* Must be able to read, understand, and sign the informed consent forms (ICF) and, when applicable, an authorization to use and disclose protected health information form (consistent with Health Insurance Portability and Accountability Act of 1996 [HIPAA] legislation as modified in 2013)
* Must be able to communicate with the investigator, and understand and comply with protocol requirements
* Must be able to wear a CG patch and perform a scan no less than once every 8 hours for the duration of the sensor periods.

Exclusion Criteria:

* Subjects who plan to use antibiotic, antifungal, antiparasitic, or antiviral treatment during the study
* Subjects using a proton pump inhibitor must be on a stable dose that will be maintained throughout the study period
* Subjects who plan to travel outside the United States during the projected study period
* Subjects who have received an experimental drug within 30 days prior to study entry
* Subjects with known milk, peanut, or tree nut allergies
* Subjects who have been diagnosed with a sexually transmitted disease including, but not limited to, HIV, syphilis, herpes, gonorrhea, hepatitis A, hepatitis B, and hepatitis C
* History of any surgery on the gastrointestinal tract except appendectomy and cholecystectomy
* Subjects with any condition that the investigator deems as a sound reason for disqualification from enrollment into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-04-29 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Technical Officer, PhD, Principal Investigator — Pendulum Therapeutics
Locations (1):
- Pendulum Therapeutics Inc, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roux de Bezieux H, Bullard J, Kolterman O, Souza M, Perraudeau F. Medical Food Assessment Using a Smartphone App With Continuous Glucose Monitoring Sensors: Proof-of-Concept Study. JMIR Form Res. 2021 Mar 4;5(3):e20175. doi: 10.2196/20175. PMID 33661120

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment through local biotechnology community network over the time period of 3/15/18-3/16/18.
Groups:
- WB-011 / Placebo: 3 capsules administered twice daily with morning and evening meal. Continuous Glucose Monitor: Abbott Freestyle Libre(™) Glucose Sensors were used throughout the study.
  Each period lasted two weeks, separated by a washout period of no-less than 3 days.
  First period - WB-011: WB-011 medical food product. Second period - Placebo: Placebo Capsules identical to those containing WB-011.
- Placebo / WB-011: 3 capsules administered twice daily with morning and evening meal. Continuous Glucose Monitor: Abbott Freestyle Libre(™) Glucose Sensors were used throughout the study.
  Each period lasted two weeks, separated by a washout period of no-less than 3 days.
  First period - Placebo: Placebo Capsules identical to those containing WB-011. Second period - WB-011: WB-011 medical food product.
Period: First Intervention
Arm/Group | WB-011 / Placebo | Placebo / WB-011
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: Washout
Arm/Group | WB-011 / Placebo | Placebo / WB-011
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | WB-011 / Placebo | Placebo / WB-011
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WB-011 / Placebo | Placebo / WB-011 | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Temperature as a Source of Unwanted Variation When Using Freestyle Libre Glucose Sensors
Description: Temperature impacts the glucose level recorded by the Freestyle Libre glucose sensors. The thermostat of the Freestyle Libre glucose sensors can be assessed.
Time Frame: Through study completion, an average of 5 weeks
Population: Technical problems with measurement of temperature data resulting in unreliable data that were uninterpretable. Therefore the endpoint was dropped.
Arm/Group | WB-011 | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: 2-hour Interstitial Glucose Area Under the Curve (AUC)
Description: Change in area under interstitial glucose concentration versus time curve (AUC) during standardized self-administered 2-hour Meal Tolerance Test.
Time Frame: Change from baseline to 2 weeks
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: min * mg/dL
Groups:
- WB-011: Participants who received the WB-011 product during either the first or second period.
- Placebo: Participants who received the placebo product during either the first or second period.
Arm/Group | WB-011 | Placebo
Number analyzed (Participants) | 6 | 6
min * mg/dL | 118.2167 (1334.929) | 613.3667 (604.2183)
Statistical Analysis 1: Comparison: WB-011 vs Placebo; Test type: Superiority; p = 0.21875, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Body Mass
Description: Weight measured via Scale
Time Frame: Change from baseline to 2 weeks
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | WB-011 | Placebo
Number analyzed (Participants) | 6 | 5
kilograms | -0.2 (2.131666) | -1.72 (2.138224)
Statistical Analysis 1: Comparison: WB-011 vs Placebo; Test type: Superiority; p = 0.90625, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Fecal Quantitative PCR Measures of Probiotic Strain Concentration
Description: Fecal quantitative PCR of product strain will be measured throughout the study if subject provide stool samples. Mass Fraction is measured and the delta between the start and end of each period is computed.
Time Frame: Change from baseline to 2 weeks
Population: Intent to treat; one subject did not provide stool samples.
Measure: Mean (Standard Deviation); unit: ng / ng
Arm/Group | WB-011 | Placebo
Number analyzed (Participants) | 5 | 5
ng / ng
  Akkermansia muciniphila | 0.0000143 (0.0000102) | -0.00000194 (0.00000367)
  Bifidobacterium infantis | 0.0000220 (0.0000259) | -0.00000286 (0.00000639)
  Clostridium beijerinckii | 0 (0) | 0 (0)
  Clostridium butyricum | 0.0000000313 (0.00000100) | -0.00000131 (0.00000294)
  Anaerobutyricum hallii | 0.000371 (0.000585) | -0.000118 (0.000230)
Statistical Analysis 1: Comparison: WB-011 vs Placebo; Paired t-test for the species Akkermansia Munciphilae; Test type: Superiority; p = 0.020, t-test, 1 sided
Statistical Analysis 2: Comparison: WB-011 vs Placebo; Paired t-test for the species Bifidobacterium infantis; Test type: Superiority; p = 0.078, t-test, 1 sided
Statistical Analysis 3: Comparison: WB-011 vs Placebo; Paired t-test for the species Clostridium beijerinckii; Test type: Superiority; No statistical test was conducted since Clostridium beijerinckii was not detected in any sample
Statistical Analysis 4: Comparison: WB-011 vs Placebo; Paired t-test for the species Clostridium butyricum; Test type: Superiority; p = 0.20, t-test, 1 sided
Statistical Analysis 5: Comparison: WB-011 vs Placebo; Paired t-test for the species Anaerobutyricum hallii; Test type: Superiority; p = 0.12, t-test, 1 sided

5. Secondary Outcome: Expected Lifespan of Continuous Glucose Monitoring (CGM) Sensors
Description: To measure the lifespan of CGM sensors, we recorded how many sensors were worn per participant during the study. Sensors were replaced either at the end of the recommended 10-day period, or when they were accidentally removed.
Time Frame: Through study completion, an average of 5 weeks
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: Number of sensors
Groups:
- All Study Participants: All participants accross all periods.
Arm/Group | All Study Participants
Number analyzed (Participants) | 6
Number of sensors | 3 (0)
Statistical Analysis 1: Comparison: All Study Participants; Test type: Other; All participants had the same number of sensors (3) throughout the study, so no statistical analysis is conducted

6. Secondary Outcome: Number of Pictures Per Day
Description: Average number of pictures per day using the smartphone application per period, used to measure study fatigue.
Time Frame: 2 weeks, (First intervention or second intervention)
Population: All participants
Measure: Mean (Standard Deviation); unit: Average number of photos per day
Groups:
- First Intervention: The first period that all participants go through, either product or placebo.
- Second Intervention: The second period that all participants crossover and go through the other intervention arm, i.e. either product or placebo.
Arm/Group | First Intervention | Second Intervention
Number analyzed (Participants) | 6 | 6
Average number of photos per day | 5.85 (2.72) | 5.46 (2.46)
Statistical Analysis 1: Comparison: First Intervention vs Second Intervention; We test whether the average number of daily photos is greater in period 1 than in period 2; Test type: Superiority; p = 0.41, t-test, 1 sided

7. Secondary Outcome: Time Between CGM-sensor Scans
Description: Average number of hours between CGM-sensor scans using the smartphone application during the study period. The subjects were instructed to scan at least every eight hours because the CGM-sensor does not save the data after eight hours without scanning.
Time Frame: 2 weeks, (First intervention or second intervention)
Population: All participants.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | First Intervention | Second Intervention
Number analyzed (Participants) | 6 | 6
hours | 2.91 (1.99) | 4.53 (2.17)
Statistical Analysis 1: Comparison: First Intervention vs Second Intervention; We test whether the average time between consecutive scans is smaller in period 1 than in period 2; Test type: Superiority; p = 0.13, t-test, 1 sided

8. Secondary Outcome: CGM-Smartphone Usability Feedback
Description: Questionnaire to assess usability of the CGM-sensor using the smartphone application.
  Question was:
  "Would you recommend others to a study like this? On a scale of 1-10 with 1 being no and 10 being absolutely"
Time Frame: Through study completion, an average of 5 weeks.
Population: Two participants did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- All Participants: Questionnaire was conducted before unblinding and focused on usability of both arms.
Arm/Group | All Participants
Number analyzed (Participants) | 4
Units on a scale | 8.25 (1.258306)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 5 weeks
Description: Used clinicaltrials.gov definitions
Arm/Group | WB-011 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT04424888/Prot_SAP_000.pdf